CLINICAL TRIAL: NCT02803073
Title: Effect of Testosterone Replacement on Exercise Capacity in Hypogonadal Men After A Recent Myocardial Infarction.
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Subjects could not be recruited
Sponsor: Texas Tech University Health Sciences Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: L16-116
Record Dates: First submitted 2016-06-08; First posted 2016-06-16 (Estimated); Last update posted 2019-11-21 (Actual); Status verified 2019-11

CONDITIONS: Hypogonadism; Acute Myocardial Infarction: Rehabilitation Phase
MeSH Terms: conditions — Hypogonadism | interventions — Testosterone; testosterone 17 beta-cypionate; Saline Solution; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Testosterone Replacement (Experimental): The experimental group will receive 0.5 ml (100 mg) testosterone cypionate Intramuscular injections each week for 11 weeks.
  Interventions: Drug: Testosterone
- Control (Placebo Comparator): Patients in the control group will receive intramuscular normal saline injections.
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Drug: Testosterone — Testosterone Cypionate Intramuscular injections will be administered weekly
  Other Names: testosterone cypionate
  Arms: Testosterone Replacement
Drug: Normal Saline — Normal Saline Intramuscular injections will be administered weekly
  Other Names: Saline
  Arms: Control

SUMMARY:
The purpose of this study is to determine the effects of testosterone replacement in hypogonadal men on exercise tolerance and cardiac rehabilitation after an acute myocardial infarction.

DETAILED DESCRIPTION:
Testosterone deficiency can decrease muscle strength. The researchers will replace testosterone in hypogonadal men undergoing rehabilitation exercises after heart attack.

ELIGIBILITY:
Inclusion Criteria:

1. All men status-post Myocardial Infarction or Non-ST Elevation-Acute Coronary Syndrome within the last 3-8 weeks enrolling in the cardiac rehabilitation program at Mission Fitness-Medical Center Hospital.
2. Baseline free testosterone levels less than age-specific normal values.
3. Males 18 years and older

Exclusion Criteria:

1. Prostate Specific Antigen greater than age based, ethnic-specific cut points (see Appendix), history of metastatic prostate cancer or symptoms suggestive of severe Benign Prostatic Enlargement.
2. Current use of testosterone, clomiphene or over the counter testosterone boosters
3. Patients initiating cardiac rehabilitation 8+ weeks after MI or Non-ST Elevation-Acute Coronary Syndrome
4. Congestive heart failure, New York Heart Association class IV
5. Life expectancy less than 1 year,
6. Baseline hematocrit of >50%
7. Allergic reactions to testosterone or testosterone vehicle (i.e. cotton seed oil, etc.)
8. Physical inability to participate in rehabilitation program (examples: severe claudication, massive obesity, etc.)
9. Participation in any other concurrent clinical trial, use of an investigational agent or therapeutic regimen within 30 days of study
10. Patients formerly diagnosed with obstructive sleep apnea.
11. Patients using opiate analgesics
12. Patients with aspartate aminotransferase/alanine aminotransferase values more than 3 times normal
13. History of Deep venous thrombosis

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Metabolic Equivalent | 12 weeks

SECONDARY OUTCOMES:
6 minute walk test | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Osama Mukarram, MD, Principal Investigator — Texas Tech University Health Sciences Center; Craig W Spellman, DO, Principal Investigator — Texas Tech University Health Sciences Center; Sandeep Dhindsa, MD, Principal Investigator — Texas Tech University Health Sciences Center
Locations (1):
- Mission Fitness-Medical Center Hospital, Odessa, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided